CLINICAL TRIAL: NCT00601367
Title: A Twenty-Eight Week, Open-Label, Safety Study of Flibanserin 50 Mgs to 100 Mgs Daily in Premenopausal European Women With HSDD
Brief Title: Flibanserin Evaluation Over 28 Additional Weeks in Hypoactive Sexual Desire Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sprout Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 511.118
Record Dates: First submitted 2008-01-15; First posted 2008-01-28 (Estimated); Results first posted 2014-06-20 (Estimated); Last update posted 2014-06-20 (Estimated); Status verified 2014-05

CONDITIONS: Sexual Dysfunctions, Psychological
MeSH Terms: conditions — Sexual Dysfunctions, Psychological

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- flibanserin flexible dose (Experimental): Initial dosage:
  Patients were to take one 50 mg flibanserin tablet in the evening.
  Subsequent dosage titrations:
  Flibanserin may have been titrated to 25 mg flibanserin b.i.d at Week 1 (Visit 2) for safety/tolerability ONLY, as determined by the clinician and given feedback from the patient.
  Flibanserin may have been up-titrated (higher daily dose) at week 4 (Visit 3) if efficacy was unsatisfactory or later in the study at a scheduled face-to-face office visit ONLY.
  Flibanserin may have been down-titrated (lower daily dose or b.i.d. regimen) at week 4 (visit 3) for safety/tolerability or later in the study at any time following patient contact with the site.
  Interventions: Drug: flibanserin flexible dose

INTERVENTIONS:
Drug: flibanserin flexible dose — Initial dosage:
  Patients were to take one 50 mg flibanserin tablet in the evening.
  Subsequent dosage titrations:
  Flibanserin may have been titrated to 25 mg flibanserin b.i.d at Week 1 (Visit 2) for safety/tolerability ONLY, as determined by the clinician and given feedback from the patient.
  Flibanserin may have been up-titrated (higher daily dose) at week 4 (Visit 3) if efficacy was unsatisfactory or later in the study at a scheduled face-to-face office visit ONLY.
  Flibanserin may have been down-titrated (lower daily dose or b.i.d. regimen) at week 4 (visit 3) for safety/tolerability or later in the study at any time following patient contact with the site.

SUMMARY:
Safety profile of flibanserin over 28 additional weeks Distribution of preferred dose regimens

ELIGIBILITY:
Inclusion Criteria:

* Women with a primary diagnosis of HSDD who still needs to be treated according to the investigator's opinion and willing to continue in this study. This continuation requires adequate compliance, in the Investigators judgement, with trial medication and the trial visit required in the parent clinical trial (Visit 1 to visit 9).
* Patients must have used a medically acceptable method of contraception [i.e., double barrier method (e.g., diaphragm or condom and spermicide), hormonal therapy (subcutaneous, injectable, intra-vaginal, or oral contraceptive), intrauterine device, tubal sterilization, or partner's surgical sterilization] for at least 3 months before the Screen Visit and continue to use that medically acceptable method of contraception during the trial.

Exclusion Criteria:

* Patients with a history of MDD within 6 months prior the Screen Visit or a score of 14 on the Beck Depression Inventory II, or a history of suicide attempt according to the Beck Scale for Suicide Ideation, or patient with any non-zero statement in the first five items for the Beck Scale for Suicide Ideation.
* Patients must have a clinically acceptable Pap smear as read by a cytology facility (no evidence of malignancy or squamous intraepithelial lesions) within 6 months before the Inclusion Visit.
* Patients with findings at the Screen Visit of pelvic inflammatory disease, urinary tract or vaginal infection/vaginitis, cervicitis, interstitial cystitis, vulvodynia, or significant vaginal atrophy.
* Patients experiencing major life stress (including parenting pressure, eldercare, loss of income, death of a family member, etc.) or relationship discord that could interfere with sexual activity, except distress about HSDD.
* Clinically significant ECG abnormalities at the Screen Visit, according to the investigators opinion or the cardiologist who have performed the ECG. The following ECG values are considered to be exclusionary: QTc intervals >480 milliseconds (ms), PR intervals >240 ms, and QRS intervals >110 ms.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Actual)
Dates: Start 2008-01; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sprout Pharmaceuticals, Study Chair — Sprout Pharmaceuticals
Locations (68):
- Austria (4):
  - 511.118.43005 Boehringer Ingelheim Investigational Site, Innsbruck
  - 511.118.43002 Boehringer Ingelheim Investigational Site, Vienna
  - 511.118.43004 Boehringer Ingelheim Investigational Site, Vienna
  - 511.118.43006 Boehringer Ingelheim Investigational Site, Wörgl
- Belgium (5):
  - 511.118.32004 Boehringer Ingelheim Investigational Site, Braine-l'Alleud
  - 511.118.32003 Boehringer Ingelheim Investigational Site, Edegem
  - 511.118.32005 Boehringer Ingelheim Investigational Site, Ghent
  - 511.118.32006 Boehringer Ingelheim Investigational Site, Hasselt
  - 511.118.32002 Boehringer Ingelheim Investigational Site, Yvoir
- Czechia (4):
  - 511.118.42001 Boehringer Ingelheim Investigational Site, Olomouc
  - 511.118.42002 Boehringer Ingelheim Investigational Site, Prague
  - 511.118.42003 Boehringer Ingelheim Investigational Site, Prague
  - 511.118.42004 Boehringer Ingelheim Investigational Site, Vřesina
- Finland (5):
  - 511.118.35801 Boehringer Ingelheim Investigational Site, Espoo
  - 511.118.35805 Boehringer Ingelheim Investigational Site, Helsinki
  - 511.118.35802 Boehringer Ingelheim Investigational Site, Oulu
  - 511.118.35803 Boehringer Ingelheim Investigational Site, Seinäjoki
  - 511.118.35804 Boehringer Ingelheim Investigational Site, Tampere
- France (11):
  - 511.118.3308A Boehringer Ingelheim Investigational Site, Blanquefort
  - 511.118.3301A Boehringer Ingelheim Investigational Site, Bordeaux
  - 511.118.3305A Boehringer Ingelheim Investigational Site, La Rochelle
  - 511.118.3314A Boehringer Ingelheim Investigational Site, Lille
  - 511.118.3314B Cabinet médical, Lille
  - 511.118.3303A Boehringer Ingelheim Investigational Site, Marseille
  - 511.118.3310A Boehringer Ingelheim Investigational Site, Marseille
  - 511.118.3312A Boehringer Ingelheim Investigational Site, Marseille
  - 511.118.3315A Cabinet Médical, Rennes
  - 511.118.3306A Boehringer Ingelheim Investigational Site, Saint-Émilion
  - 511.118.3311A Boehringer Ingelheim Investigational Site, Toulouse
- Germany (7):
  - 511.118.49004 Boehringer Ingelheim Investigational Site, Berlin
  - 511.118.49001 Boehringer Ingelheim Investigational Site, Bonn
  - 511.118.49006 Boehringer Ingelheim Investigational Site, Dresden
  - 511.118.49008 Boehringer Ingelheim Investigational Site, Frankfurt
  - 511.118.49003 Boehringer Ingelheim Investigational Site, Freiburg im Breisgau
  - 511.118.49002 Boehringer Ingelheim Investigational Site, Hanover
  - 511.118.49005 Boehringer Ingelheim Investigational Site, Leipzig
- Hungary (4):
  - 511.118.36001 Boehringer Ingelheim Investigational Site, Budapest
  - 511.118.36005 Boehringer Ingelheim Investigational Site, Kecskemét
  - 511.118.36003 Boehringer Ingelheim Investigational Site, Szeged
  - 511.118.36004 Boehringer Ingelheim Investigational Site, Szentes
- Italy (3):
  - 511.118.39004 Boehringer Ingelheim Investigational Site, Catania
  - 511.118.39001 Boehringer Ingelheim Investigational Site, Pavia
  - 511.118.39003 Boehringer Ingelheim Investigational Site, Torino
- Netherlands (7):
  - 511.118.31006 Boehringer Ingelheim Investigational Site, Almere Stad
  - 511.118.31001 Boehringer Ingelheim Investigational Site, Amsterdam
  - 511.118.31004 Boehringer Ingelheim Investigational Site, Apeldoorn
  - 511.118.31003 Boehringer Ingelheim Investigational Site, Bilthoven
  - 511.118.31007 Boehringer Ingelheim Investigational Site, Den Helder
  - 511.118.31005 Boehringer Ingelheim Investigational Site, Enschede
  - 511.118.31002 Boehringer Ingelheim Investigational Site, Nieuwegein
- Spain (4):
  - 511.118.34004 Boehringer Ingelheim Investigational Site, Barcelona
  - 511.118.34003 Boehringer Ingelheim Investigational Site, Manresa (Barcelona)
  - 511.118.34002 Boehringer Ingelheim Investigational Site, Mataró-Barcelona
  - 511.118.34001 Boehringer Ingelheim Investigational Site, Ourense
- Sweden (6):
  - 511.118.46004 Boehringer Ingelheim Investigational Site, Kungsbacka
  - 511.118.46009 Boehringer Ingelheim Investigational Site, Lund
  - 511.118.46001 Boehringer Ingelheim Investigational Site, Stockholm
  - 511.118.46006 Boehringer Ingelheim Investigational Site, Stockholm
  - 511.118.46005 Boehringer Ingelheim Investigational Site, Uppsala
  - 511.118.46003 Boehringer Ingelheim Investigational Site, Västerås
- United Kingdom (8):
  - 511.118.44009 Boehringer Ingelheim Investigational Site, Chorley
  - 511.118.44004 Boehringer Ingelheim Investigational Site, Fisherwick, Lichfield
  - 511.118.44008 Boehringer Ingelheim Investigational Site, Glasgow
  - 511.118.44003 Boehringer Ingelheim Investigational Site, Headington, Oxford
  - 511.118.44001 Boehringer Ingelheim Investigational Site, London
  - 511.118.44002 Boehringer Ingelheim Investigational Site, London
  - 511.118.44007 Boehringer Ingelheim Investigational Site, South Brent
  - 511.118.44010 Boehringer Ingelheim Investigational Site, Waterloo, Liverpool

RESULTS

PARTICIPANT FLOW:
Groups:
- Flibanserin Flexible Dose: Initial dosage:
  Patients were to take one 50 mg flibanserin tablet in the evening.
  Subsequent dosage titrations:
  Flibanserin may have been titrated to 25 mg flibanserin b.i.d at Week 1 for safety/tolerability ONLY, as determined by the clinician and given feedback from the patient. Flibanserin may have been up-titrated (higher daily dose) at week 4 if efficacy was unsatisfactory or later in the study at a scheduled face-to-face office visit ONLY. Flibanserin may have been down-titrated (lower daily dose or b.i.d. regimen) at week 4 for safety/tolerability or later in the study at any time following patient contact with the site.
Period: Overall Study
Arm/Group | Flibanserin Flexible Dose
Started | 480
Completed | 293
Not Completed | 187

BASELINE CHARACTERISTICS:
Groups:
- Flibanserin Flexible Dose: Initial dosage:
  Patients were to take one 50 mg flibanserin tablet in the evening.
  Subsequent dosage titrations:
  Flibanserin may have been titrated to 25 mg flibanserin b.i.d at Week 1for safety/tolerability ONLY, as determined by the clinician and given feedback from the patient.
  Flibanserin may have been up-titrated (higher daily dose) at week 4 if efficacy was unsatisfactory or later in the study at a scheduled face-to-face office visit ONLY. Flibanserin may have been down-titrated (lower daily dose or b.i.d. regimen) at week 4 for safety/tolerability or later in the study at any time following patient contact with the site.
  flibanserin flexible dose: Initial dosage: Patients were to take one 50 mg flibanserin tablet in the evening.
  Subsequent dosage titrations:
  Flibanserin may have been titrated to 25 mg flibanserin b.i.d at Week 1 (Visit 2) for safety/tolerability ONLY, as determined by the clinician and given feedback from the pati
Arm/Group | Flibanserin Flexible Dose
Number analyzed (Participants) | 480
Age, Customized [Number; unit: participants]
  18-29 years | 97
  30-39 years | 211
  40-49 years | 170
  50 years and older | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 480
  Male | 0
Race/Ethnicity, Customized [Number; unit: participants]
  White | 442
  White Hispanic | 8
  Black | 4
  Missing | 26

OUTCOME MEASURES:

1. Primary Outcome: Frequency of Adverse Events
Time Frame: 28 weeks
Measure: Number; unit: participants with any adverse event
Arm/Group | Flibanserin Flexible Dose
Number analyzed (Participants) | 480
participants with any adverse event
  patients with any adverse event | 331
  patients with drug-related adverse events | 206
  patients with adverse events leading to discontinu | 58
  patients with severe adverse events | 51
  patients with serious adverse events | 9

ADVERSE EVENTS:
Arm/Group | Flibanserin Flexible Dose
Serious Adverse Events (participants affected / at risk) | 9/480
Other Adverse Events (participants affected / at risk) | 275/480
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Flibanserin Flexible Dose (N=480)
gastroenteritis (Infections and infestations) | 1 (1)
Breast Cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Migraine with aura (Nervous system disorders) | 1 (1)
Neuralgia (Nervous system disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Uterine polyp (Reproductive system and breast disorders) | 2 (2)
ovarian cyst (Reproductive system and breast disorders) | 1 (1)
Exomphalos (Congenital, familial and genetic disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Flibanserin Flexible Dose (N=480)
Fatigue (Nervous system disorders) | 69 (78)
Headache (Nervous system disorders) | 51 (71)
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 47 (54)
Nausea (Gastrointestinal disorders) | 41 (47)
Dizziness (Nervous system disorders) | 40 (52)
Somnolence (Nervous system disorders) | 27 (29)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No